CLINICAL TRIAL: NCT07169643
Title: Darbepoetin in Patients Candidates for Liver Transplant: Randomized Clinical Trial Protocol. (EPO-LT Trial)
Brief Title: Darbepoetin in Patients Candidates for Liver Transplant. (EPO-LT Trial)
Acronym: EPO-LT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPO-LT Trial
Record Dates: First submitted 2025-08-24; First posted 2025-09-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant; Complications
Keywords: living kidney trasplant
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: This is a phase III, multicenter, randomized clinical trial to evaluate the the efficacy and safety of DP administration in patients on the liver transplant waiting list to reduce intraoperative red blood cell concentrate transfusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Darbepoetin arm (Experimental): Darbepoetin (DP) 1.5 mcg/kgsub cutaneously, monthly (The patients will receive medication monthly until the liver transplant is performed or if it has not yet been transplanted, a maximum of 3 doses)
  Interventions: Drug: Darbepoetin (DP)
- No intervention arm (No Intervention): No administration darbepoetin(DP).

INTERVENTIONS:
Drug: Darbepoetin (DP) — Darbepoetin (DP) 1.5 mcg/kg subcutaneously, monthly (The patients will receive medication monthly until the liver transplant is performed or if it has not yet been transplanted, a maximum of 3 doses)
  Arms: Darbepoetin arm

SUMMARY:
This is a national multicenter, randomized clinical trial to evaluate the the efficacy and safety of DP administration in patients on the liver transplant waiting list to reduce intraoperative red blood cell concentrate transfusion.

DETAILED DESCRIPTION:
Patients will be randomized to receive (1:1):

1. Intervention group: Darbepoetin (DP) 1.5 mcg/kg subcutaneously, monthly (The patients will receive medication monthly until the liver transplant is performed or if it has not yet been transplanted, a maximum of 3 doses)
2. Control group: Do not Darbepoetin All patients will be evaluated to rule out vitamin B12 and folic acid deficiencies, and supplementation with 1000 mcg/day and 10 mg/day, respectively, will be provided if necessary. All patients, on the liver transplant list, will receive ferric carboxymaltose 1000 mg IV (every month) according to standard clinical practice Patients will be followed for 3 months after LT

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients on the official liver transplant waiting list
3. Hemoglobin (Hb) level ≤ 11.5 g/dL
4. Women of child-bearing potential* must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence** (only if refraining from heterosexual intercourse during the period of twelve months). Hormonal contraceptive methods will be avoided due to the risk of adverse events and impairment of liver function.

   * A woman will be considered of childbearing potential, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as 0 menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single follicle stimulating hormone measurement is insufficient. ** Sexual abstinence should only be used as a contraceptive method if it is in line with the subjects' usual and preferred lifestyle. Periodic abstinence (calendar, symptothermal, post ovulation methods) is not an acceptable method of contraception.

Exclusion Criteria:

* 1. Acute/subacute liver failure (see appendix 7) 2. Patients with acute-on-chronic liver failure grade III and/or MELD > 35 3. History of thrombosis, including portal vein thrombosis 4. Significant coronary artery disease (requiring angioplasty and/or coronary stent) 5. Serum ferritin > 800 ng/mL and SAT > 50% 6. Anticoagulant/antiplatelet therapy 7. History of seizures 8. Uncontrolled hypertension (requiring ≥2 antihypertensive drugs) 9. Active infection/sepsis (see appendix 8) 10. Lack of patient consent. 11. Pregnancy or breastfeeding. 12. Patients included in other clinical trials in the month before inclusion. 13. Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
to investigate the efficacy and safety of darbepoetin (DP) administration in patients on the liver transplant (LT) waiting list to reduce intraoperative red blood cell concentrate transfusion. | perioperative
  Difference in the percentage of patients receiving intraoperative (LT) red blood cell transfusions between the intervention group and the control group.

SECONDARY OUTCOMES:
Investigate the increase in hemoglobin levels | through study completion, an average of 1 year
  Absolute differences from baseline in hemoglobin levels basal and at 4, 8, 12 or 16 weeks after the administration of DP, or at the time of liver transplantation, between the intervention group and the control group
Investigate the difference in the percentage of patients receiving intraoperative and during the first 24h after LT, red blood cell concentrate transfusion between the intervention and control groups | baseline Visit , perioperative visit, month 3 postoperative
  Difference in the percentage of patients receiving intraoperative and during the first 24h after LT, red blood cell transfusions between the intervention group and the control group
Investigate the difference in the percentage of patients receiving intraoperative massive transfusion between the intervention and control groups. | perioperative visit
  Difference in the percentage of patients receiving massive transfusions(>6 units of red blood cells)
Investigate the difference in the percentage of patients who developed severe postoperative complications between the intervention and control groups. | Difference in the 3-month severe postoperative complications
  assessed by the Comprehensive Charlson Index, between groups
Investigate the difference in the overall cost of the transplantation from surgery to three months post-transplant, between the intervention and control groups. | three months post-transplant
  Difference in the overall cost (direct and indirect) of the transplantation, conducting a cost-effective analysis between groups
To evaluate the difference in postoperative graft survival , between groups | the 3 month, 6, and 12 months, postoperative graft survival after liver transplantation, between groups
  To evaluate the difference in the 3 month, 6, and 12 months, postoperative graft survival after liver transplantation, between groups
To investigate the difference in the 3 month, 6, and 12 months, postoperative patient survival after liver transplantation, between groups | in the 3 month, 6, and 12 months, postoperative patients survival after liver transplantation
  To evaluate the difference in the 3 month, 6, and 12 months, postoperative patients' survival after liver transplantation, between groups
Impact of DP treatment on the hemostatic profile of patients with chronic liver disease, comparing the changes in the following coagulation marker beta-TG at basal and 4 weeks after administration | at basal visit and month1
  changes in the beta-TG marker (mg/mL)
Impact of DP treatment on the changes in the PF4 profile of patients with chronic liver disease, comparing the changes in the fPF4 coagulation marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the e PF4 (heprin antibody test ) in (IU/dL)
Impact of DP treatment on the hemostatic profile of patients with chronic liver disease, comparing the fibrinogen marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the fibrinogen (g/L)
Impact of DP treatment on the hemostatic profile of patients with chronic liver disease, comparing the changes in theTM-TGA marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the TM-TGA(ng/mL)
Impact of DP treatment , comparing the changes in the following coagulation CTL marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the CLT, (clothing and lysis time test ) (minutes) between groups
Impact of DP treatment on the fibrinolitic profile of patients with chronic liver disease, comparing the changes iD dimer markers at basal and 4 weeks after administration | at basal visit and month1
  changes in the D dimer (micrograms/L) between groups
Impact of DP treatment comparing the changes in the TAT marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the TAT (trombi-antitrombin) (minutes), between groups
Impact of DP treatment comparing the changes in the heptacidin marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the hepcidin (nmol/dL), between groups
Impact of DP treatment on the erythropoietin marker at basal and 4 weeks after administration | at basal visit and month1
  changes in the erythropoietin (mU/mL) between groups
To explore the impact of anemia on complications of portal hypertension | through study completion, an average of 1 year
  the number and type of acute decompensations (acute gastrointestinal bleeding, infection,Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
To explore the impact of the anemia on the quality of life measured by the EuroQol-5D scale , in both groups. | through study completion, an average of 1 year
  the quality of life measured by the EuroQol-5D scale of quality of live european
To explore the predictors of poor response to DP treatment | base line visit, month 1, month 2, month 3, month 6.
  defined as the increase in the hemoglobin level < 1 g/dL after 1 month of treatment.
Proportion of patients and severity of treatment-related adverse events during the study period, | through study completion, an average of 1 year
  Proportion of patients and severity of treatment-related adverse events during the study period,

CONTACTS AND LOCATIONS:
Overall Officials: Annabel Blasi, Dr, Principal Investigator — Fundació de Recerca Clínic Barcelona - Institut D'Investigacions Biomèdiques Agustí Pí i Sunyer
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No